CLINICAL TRIAL: NCT00173654
Title: Mutation Analysis of 17βhydroxysteroid Dehydrogenase 3 Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700825
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2005-08

CONDITIONS: Pseudohermaphroditism
MeSH Terms: conditions — Disorders of Sex Development | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: blood drawing

SUMMARY:
To disclose the molecular pathology of our 3 families with 17βHSD3 deficiency.

DETAILED DESCRIPTION:
17βhydroxysteroid dehydrogenase 3 (17βHSD3) deficiency is a rare cause of male pseudohermaphroditism. The incidence is reported to be 1: 147,000 in the Netherlands. Fewer than one hundred affected 46, XY males were reported in the literature, and no such case has been reported in Taiwan before. The 46, XY patients have ambiguious or complete female external genitalia. They are mostly unrecognized at birth and reared as female. They often draw medical attention when they receive operation for inguinal hernia or during puberty, clitoromegaly and musculization were noticed. However, the homozygous or compound heterozygous genetic females are asymptomatic. The 17βHSD3 catalyze the conversion of androstenedione to testosterone, the last step in the synthesis of testosterone. Therefore, the serum levels of androstenedione are elevated and testosterone or dihydrotestosterone are in the low range in these affected 46, XY individuals. The clinical diagnosis is made by HCG stimulation test, because androstenedione-to-testosterone ratio is abnormally elevated in these patients. But the molecular basis of 17βHSD3 deficiency was not determined till recent decade.

The HSD17B3 gene was elucidated in 1994, and composed of 11 exons. Several missence mutation and splice mutation were identified. But the precise action and tissue distribution of 17βHSD3 still need to be clarified. The Wölffian ducts virilze normally in the embryonic stage and the serum concentration of testosterone achieve to the normal range in the pubertal stage. The exact mechanism is not understood clearly and peripheral conversion under other isozymes was suggested in some studies.

The purpose of this study is to disclose the molecular pathology of our 3 families with 17βHSD3 deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 17β-hydroxysteroid dehydrogenase 3 deficiency and their family

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2005-08; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ching Tung, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan